CLINICAL TRIAL: NCT05952960
Title: Optimizing Open Label Placebo Rationales for Chronic Pain
Brief Title: Optimizing Open Label Placebo Rationales
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 196178
Record Dates: First submitted 2023-05-01; First posted 2023-07-19 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TAU Rationale (Other): Rationale based on prior OLP studies (e.g. Kaptchuk et al., 2010)
  Interventions: Other: Placebo
- Mindfulness Rationale (Other): Rationale based on mindfulness meditation
  Interventions: Other: Placebo
- Suspension of Disbelief Rationale (Other): Rationale based on suspending disbelief about the placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Open Label Placebo + Rationale

SUMMARY:
A 3-arm randomized trial where all chronic pain patients will receive honest placebos, but the information about the placebos will differ between conditions. Outcomes are measured for 21 days and a qualitative survey will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* chronic pain
* 18 years old
* English speaking
* have a smartphone or computer with video access
* Taking prescription opioids for chronic pain
* the chronic pain is concentrated into the patient's lower back.

Exclusion Criteria:

* suspect an allergy to any placebo ingredient
* problematic substance use
* cancer diagnosis causing pain
* anticipated change in opioid script during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Pain Reports | 21 days
  Brief Pain Inventory: Pain intensity and pain interference

SECONDARY OUTCOMES:
Opioids | 21 Days
  Quantity of prescription opioids taken

CONTACTS AND LOCATIONS:
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided